CLINICAL TRIAL: NCT06874088
Title: Evaluation of Clinical and Radiographic Prognosis of Pulpotomy Treatment Performed on Teeth with Different Symptoms and Stages of Root Development: a Retrospective Study
Brief Title: Clinical and Radiographic Outcomes of Pulpotomy in Teeth with Different Symptoms and Root Stages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammed Alagöz (Other)
Responsible Party: Sponsor-Investigator, Muhammed Alagöz, research assistant, Ataturk University
Organization: Ataturk University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/13; atatürk üniversitesi (Other: Atatürk Üniversitesi Diş Hekimliği Fakültesi)
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Reversible Pulpitis; Irreversible Pulpitis; Mature Teeth; Immature Teeth
Keywords: Vital pulp therapy; Pulpotomy; Dentin bridge formation; Periapical Index; Retrospective study
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pulpotomy (Experimental): In cases where pulp exposure exceeded 2 mm, the pulpotomy procedure was performed. The intervention commenced with the excision of the pulp chamber roof using a steel round bur. The coronal pulp tissue was then amputated at the level of the canal orifices utilizing a sterile sharp spoon excavator. Hemostasis was achieved by applying a sterile cotton pellet moistened with physiological saline for 3-5 minutes. Once hemostasis was confirmed, the cavity was further disinfected with 2.5% sodium hypochlorite. Subsequently, a 2 mm thick layer of mineral trioxide aggregate was placed over the pulp stump and covered with a resin-modified glass ionomer cement. To enhance adhesion, the cavity walls were conditioned with 35% orthophosphoric acid following the removal of residual material using a steel round bur. After the application of a dentin bonding agent, the definitive restoration was completed with composite resin using an incremental layering technique.
  Interventions: Procedure: Pulpotomy with Calcium Silicate-Based Bioceramics in Permanent Teeth

INTERVENTIONS:
Procedure: Pulpotomy with Calcium Silicate-Based Bioceramics in Permanent Teeth — This intervention involves performing pulpotomy using calcium silicate-based bioceramic materials, MTA and Biodentine™, in both mature and immature permanent teeth diagnosed with reversible or irreversible pulpitis. The study uniquely evaluates the long-term clinical and radiographic success of these materials by assessing pulp healing, dentin bridge formation, and periapical healing over a 24-month follow-up period. Additionally, this study compares clinical survival rates between mature and immature teeth, contributing to the growing body of evidence on the efficacy of pulpotomy in cases traditionally considered for root canal treatment. Unlike conventional pulpotomy studies, this research incorporates retrospective data analysis to align with international standards, addressing gaps in existing literature.

SUMMARY:
Pulpotomy is a vital pulp therapy (VPT) method used to maintain pulp vitality by removing inflamed or infected coronal pulp tissue while preserving the health and function of radicular pulp. This procedure supports root development in young permanent teeth and helps prevent long-term complications associated with apexogenesis.

Recent studies indicate that pulpotomy can achieve success rates exceeding 90%, even in cases of symptomatic irreversible pulpitis, challenging traditional contraindications. Notably, this high success rate has been observed in both immature and mature permanent teeth, expanding the applicability of pulpotomy across different developmental stages.

Modern materials such as Mineral Trioxide Aggregate (MTA) and Biodentine™ have been widely adopted in regenerative dentistry due to their biocompatibility and superior sealing properties. These materials are used effectively in both immature and mature teeth, contributing to the long-term success of vital pulp therapy.

DETAILED DESCRIPTION:
This retrospective study evaluates the effectiveness of bioceramic materials such as Mineral Trioxide Aggregate (MTA) and Biodentine™ in the treatment of both reversible and irreversible pulpitis cases. The study compares the clinical survival rates of pulpotomy in teeth with mature and immature root structures and assesses long-term biological outcomes, including pulp healing, dentin bridge formation, and periapical healing. Additionally, the study aims to address gaps in the literature by providing retrospective data from our country and making it comparable with international standards.

Detailed Description

Study Objectives

To retrospectively analyze the effectiveness of bioceramic materials such as MTA and Biodentine™ in cases of reversible and irreversible pulpitis.

To compare the clinical survival rates of pulpotomy in teeth with mature and immature root structures.

To evaluate long-term biological outcomes based on criteria such as pulp healing, dentin bridge formation, and periapical healing.

To provide retrospective data from our country that can be compared with international standards, addressing gaps in the existing literature.

Clinical Procedure

The treatment protocol was performed by a single pediatric dentist. After local anesthesia, rubber dam isolation was applied to enhance visibility and maintain asepsis. The enamel, dentin, and pulp chamber roof were sequentially removed using ISO 021-023 diamond and steel round burs (NTI-Kahla GmbH, Kahla, Germany). The coronal pulp tissue was amputated up to the root canal orifices using a sterile sharp steel round bur. Hemostasis was achieved by applying a sterile cotton pellet soaked in 2.5% sodium hypochlorite and saline solution.

Following hemostasis, the bioceramic materials were freshly mixed according to the manufacturer's recommendations. A 2-3 mm thick layer of either MTA (Biofactor, Imicryl Dental, Konya, Turkey) or Biodentine™ (Septodont, France) was carefully applied to the pulp chamber floor. The material was then covered with a resin-modified glass ionomer cement (Ionoseal, VOCO GmbH, Cuxhaven, Germany). Any excess material adhering to the cavity walls was removed using a steel round bur to ensure optimal adhesion of the restorative material and to prevent microleakage. The cavity walls were then etched with 35% orthophosphoric acid (Vococid, Voco, Germany), followed by the application of a dentin bonding agent (Futurabond-U, Voco, Germany). The final restoration was completed using a composite resin (Solare-X, GC, Tokyo, Japan) in a layering technique. Occlusal adjustments and polishing were performed in the same session.

Follow-up and Outcome Evaluation

Clinical and radiographic follow-up evaluations were conducted at an average of 24 months post-treatment. Clinical parameters such as spontaneous pain, nocturnal pain, vestibular swelling, pathological mobility, and percussion or palpation sensitivity were recorded before and after treatment to assess success.

Radiographic evaluations were performed using the Periapical Index (PAI) to assess periapical healing, and the presence of a dentin bridge was also examined in follow-up radiographs. Additionally, root development was assessed using the Moorrees Index in initial and follow-up radiographs.

This study provides valuable insight into the long-term effectiveness of pulpotomy in mature and immature teeth, contributing to the existing body of knowledge on vital pulp therapy.

ELIGIBILITY:
Inclusion Criteria:

* Mature and immature permanent teeth exposed to caries.
* Teeth with reversible or irreversible clinical symptoms.
* Periapical index (PAI) scores of 1 or 2 (indicating healthy or mildly inflamed periapical tissues) at baseline.
* Patients without any systemic disorders.

Exclusion Criteria:

* Radiographic evidence of periradicular or interradicular lesions.
* Presence of internal or external root resorption.
* Patients with systemic conditions that may compromise healing, such as diabetes or immunosuppression.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Clinical Success of Pulpotomy in Mature and Immature Permanent Teeth | 24 months
  Clinical success was determined based on the absence of symptoms such as spontaneous pain, tenderness to percussion, swelling, sinus tract formation, and abnormal mobility. Teeth exhibiting normal function without signs of pulpal or periapical pathology during follow-up examinations were classified as clinically successful. Additionally, patient-reported outcomes, including the resolution of preoperative symptoms and continued functionality, were considered in the clinical assessment.
Radiographic Success of Pulpotomy in Mature and Immature Permanent Teeth | 24 months
  Radiographic success was defined by the absence of periapical radiolucency, internal or external root resorption, and signs of pathological changes in the periradicular tissues. Teeth demonstrating a well-preserved root structure, maintained pulp space dimensions, and no evidence of progressive pathology on follow-up radiographs were considered radiographically successful. Consistent findings across multiple follow-up intervals further confirmed the stability of pulpal and periapical health post-pulpotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Dentistry, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided